CLINICAL TRIAL: NCT02271516
Title: A Phase I, Open-label, Dose-escalation Study to Determine the Maximum Tolerance Dose (MTD) and to Evaluate the Safety of 188Re-BMEDA-liposome in Patient With Primary Solid Tumor in Advanced or Metastatic Stage.
Brief Title: to evaluate188Re-BMEDA-liposome in Patient With Primary Solid Tumor in Advanced or Metastatic Stage
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Some concerns arose for the accumulation of radioactivity in liver and spleen.
Sponsor: National Atomic Research Institute, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QCR12009
Record Dates: First submitted 2014-10-15; First posted 2014-10-22 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 188Re-BMEDA-liposome (Experimental): Stage I:
  188Re-BMEDA-liposomes, 14±1.4 mCi, single dose
  Stage II:
  188Re-BMEDA-liposomes, dose-escalation, single dose Dose Level Dose of 188Re-BMEDA-liposome (mCi/kg)
  1. 0.42±0.04 mCi/kg
  2. 0.63±0.06 mCi/kg
  3. 0.84±0.08 mCi/kg
  4. 1.05±0.11 mCi/kg
  5. 1.26±0.13 mCi/kg
  6. 1.47±0.15 mCi/kg
  Interventions: Radiation: 188Re-BMEDA-liposome

INTERVENTIONS:
Radiation: 188Re-BMEDA-liposome — EKG at baseline and in 24hours after administration

SUMMARY:
This is a study to determine the maximum tolerance dose (MTD) and to evaluate the safety of 188Re-BMEDA-liposome in patient with primary solid tumor in advanced or metastatic stage.

DETAILED DESCRIPTION:
Rhenium-188 is an ideal radionuclide for therapeutic use due to its maximum beta emission of 2.12MeV, short physical half-life of 16.9 hours, and its 155-keV gamma emission for imaging purposes. 188Re-BMEDA-liposome consists of 2 separate components (Rhenium-188 and liposome) and BMEDA as a linker. This study aims to find the MTD, evaluate the safety, efficacy profiles and investigate the biodistribution, radioactivity and radiation dosimetry of 188Re-BMEDA-liposome on primary solid tumor in metastatic stage patient by a single intravenous injection course.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically confirmed diagnosis of primary solid tumor, and with pathologically or radiologically documented metastases
* Disease that is measurable or evaluable by RECIST 1.1 criteria (for Solid Tumors)
* Patient with metastatic cancer that are refractory to current standard/available therapies

Exclusion Criteria:

* brain metastases
* serious concurrent infection or nonmalignant illness that is uncontrolled
* uncontrolled intercurrent illness
* Immunocompromised
* significant traumatic injury within 3 weeks before Day 0
* History of hypersensitivity to any component of study drug

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Determine the MTD | up to 30 days per cohort
  The design will use cohort of 3 patients. If none of the first 3 patients experience DLT, then dose escalation will proceed for the next dose level of patients unless the present dose level is level 6 (1.47±0.15 mCi/kg).

SECONDARY OUTCOMES:
change in vital signs and pysical examination | from day 0 to up t0 60 days per cohort
  assess the safety issue from the change in vital signs (BP, PR, RR and temperature) and physical examinations
change in lab data | from day 0 to up t0 60 days per cohort
  assess the safety issue from the change in lab data including heatology lab data change, Biochemistry laboratory data change and urinalysis data change
Adverse event(s) | from day 0 to up t0 60 days per cohort
  assessed by NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) v4.03
Serious Adverse event(s) | from day 0 to up t0 60 days per cohort
  All AE(s) and SAE(s) which occurred within follow-up visit after the single dose administration of study drug should be followed until resolution or the event is considered stable.
Change in EKG | in 24hrs
  Patient will be examined the EKG by standard 12-lead at screen visit for eligibility. After enrollment, patient will be attached on a 24h-portable EKG monitor to monitoring EKG before and post-administration of Stage I and II low dose and therapeutic infusion dose for 24hrs

CONTACTS AND LOCATIONS:
Overall Officials: Shyh-Jen Wang, MD, Principal Investigator — Taipei Veterans General Hospital (Taiwain)
Locations (1):
- Taipei Veterans General Hospital (Taiwain), Taipei, Taiwan